CLINICAL TRIAL: NCT06969105
Title: A Randomized Controlled Trial of Music Use in Parturients Admitted to Labor & Delivery
Brief Title: Music Use in Parturients Admitted to Labor & Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005897
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Pain; Patient Satisfaction
Keywords: music; labor and delivery; parturients; anxiety; analgesia; anesthesia; pain; epidural
MeSH Terms: conditions — Anxiety Disorders; Pain; Patient Satisfaction; Agnosia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: One group will listen to music (intervention) and the other group will not listen to music (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): Subjects randomized to this arm will listen to music for a 10 minute duration.
  Interventions: Other: Music
- Control Group (No Intervention): Subjects randomized to this arm will not listen to music for a 10 minute duration.

INTERVENTIONS:
Other: Music — Prior to randomization, all participants will pre-select their preferred music genre. If randomized to the music group, their preferred music genre will be played for a 10 minute duration.
  Arms: Music Group

SUMMARY:
The goal of this clinical trial is to learn if music use affects anxiety or pain levels in parturients admitted to labor and delivery. It will also learn about the effect of music use on patient satisfaction. The main questions it aims to answer are:

Does music use affect anxiety levels in parturients admitted to labor and delivery? Does music use affect pain levels in parturients admitted to labor and delivery? Does music use affect patient satisfaction in parturients admitted to labor and delivery?

Researchers will compare music to a control (no music) to see if music affects anxiety levels in parturients admitted to labor and delivery.

Participants will:

Listen to music or listen to no music for a 10 minute duration in the labor and delivery unit.

Answer questions about anxiety and pain levels at a few different timepoints. Have information collected from medical charts (vital signs and cervical dilation).

Rate their satisfaction with care.

DETAILED DESCRIPTION:
Subjects will be asked their preferred music choice before they are randomly assigned to either the intervention music group, or the no music control group.

The study's active intervention group will be listening to the subject's preferred music for a duration of 10 minutes. The subjects will listen to their preferred music choice played from a speaker connected to an audio device, both supplied by the research team. The investigator and the patient will collaborate on patient positioning of the audio device for sound to optimize comfort and safety during the study intervention. Researchers will confirm the volume of the music and assess subject's comfort before leaving the room for 10 minutes while they listen to music. Subjects must turn off all other noises such as television, other music being played, phone calls ringer/vibration, and texting notifications will be turned off prior to initiation of the study. Phone calls and texting may be left on for subject's who request this. The study team will wait outside the door for 10 minutes, before re-entering. Nursing and providers essential to care will be notified that the subject is participating in the study to ensure no one enters the room unless medically necessary or in case of emergency during this 10-minute time period.

The Control group will not listen to music. The study team will still leave the room for 10 minutes and then re-enter to continue collecting data at each of the time points as below:

Before the intervention begins, researchers will collect from all parturient subjects' their anxiety score (on a scale of 0-10, with 0 being no anxiety), ask them to complete the STAI questionnaires on paper to collect their scores (submitted) and pain score, and record the time data was collected. Researchers will also record clinical data from the EMR for the parturient subject or ask the nurses for the data at the time they take these readings (see Data Collection Form).

If parturient subjects request labor analgesia and have an epidural catheter placed, researchers will collect the same data from parturient subjects both at the time that the request is made and within 30 minutes of the catheter being placed. The data collected from these two timepoints is an optional component of the study (see Informed Consent Form). The subjects can consent ahead of time in the ICF but may withdraw consent for these 2 data points and still be in the rest of the study as the data collected at these 2 timepoints are secondary objectives to explore. If a member of the research team is not in the room at the time this happens, researchers will not collect Anxiety, STAI or pain score and will only collect what is available from the charts, as per the Data Collection Form.

After the intervention (or time has passed, if they are in the control group), the same information will be collected from all participants a second time (see Data Collection Form). Parturient satisfaction will be recorded (Data Collection Form). Nurses on the subject's normal care team will be asked to assist with collecting the vitals for the data collection forms.

All procedures are occurring for research purposes only. Initial vitals collected will be done as per standard care and data will only be pulled later from charts or researchers will ask the nurses for the information as they are collecting it. Later vitals collected, if done at a time where they are not being collected for standard care, will be collected for research only - by the standard care team nurses.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Laboring parturients or those scheduled for an induction of labor
* Able to provide informed consent
* American Society of Anesthesiologists (ASA) physical status rating of II-III

Exclusion Criteria:

* Patient refusal
* Impaired hearing
* Patient is taking at least one anxiolytic medication daily at baseline
* Intrauterine fetal demise
* Severe psychiatric disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline and 0 hours post-intervention
  Anxiety will be assessed in two ways. The first using a 0-10 numeric rating scale in which subjects rate their self-perceived anxiety level on this scale. Secondly, they will answer survey questions on the State-Trait Anxiety Inventory questionnaire.

SECONDARY OUTCOMES:
Pain Level | Baseline to 0 hours post-intervention
  Pain will be assessed on a 0-10 numeric rating scale in which subjects rate their self-perceived level of pain.
Patient Satisfaction | 0 hours post-intervention
  Patient satisfaction will be assessed using a survey question asking how satisfied the patient is with their care. Subject will rate their satisfaction level as very poor, somewhat poor, average, satisfied, or very satisfied.
Anxiety | Request of labor analgesia and 0,1 hour post-epidural catheter placement
  Anxiety levels will be assessed using a 0-10 numerical rating scale and on the State Trait Anxiety Inventory questionnaire. Subject will rate their self-perceived anxiety level and answer survey questions.
Pain Level | Request of labor analgesia and 0,1 hours post-epidural catheter placement
  Pain will be assessed using a 0-10 numerical rating scale. Subject will rate their self-perceived pain level on this scale.
Blood Pressure | Request of labor analgesia and 0,1 hours post-epidural catheter placement
  Blood pressure will be recorded in units of millimeters of mercury (mmHg) from an automated vital signs monitor that the patient will already be monitored on upon arrival to the unit.
Heart Rate | Request of labor analgesia and 0,1 hours post-epidural catheter placement
  Heart rate will be recorded in units of beats per minute (bpm) from an automated vital signs monitor that the patient will already be monitored on upon arrival to the unit.
Oxygen Saturation | Request of labor analgesia and 0,1 hours post-epidural catheter placement
  Oxygen saturation will be recorded as a percentage (SpO2) from an automated vital signs monitor that the patient will already be monitored on upon arrival to the unit.
Blood Pressure | Baseline to 0 hours post-intervention
  Blood pressure will be recorded in units of millimeters of mercury (mmHg) from an automated vital signs monitor that the patient will already be monitored on upon arrival to the unit.
Oxygen Saturation | Baseline to 0 hours post-intervention
  Oxygen saturation will be recorded as a percentage (SpO2) from an automated vital signs monitor that the patient will already be monitored on upon arrival to the unit.
Heart Rate | Baseline to 0 hours post-intervention
  Heart rate will be recorded in units of beats per minute (bpm) from an automated vital signs monitor that the patient will already be monitored on upon arrival to the unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tabarro CS, de Campos LB, Galli NO, Novo NF, Pereira VM. [Effect of the music in labor and newborn]. Rev Esc Enferm USP. 2010 Jun;44(2):445-52. doi: 10.1590/s0080-62342010000200029. Portuguese. PMID 20642059
- [Background] Phumdoung S, Good M. Music reduces sensation and distress of labor pain. Pain Manag Nurs. 2003 Jun;4(2):54-61. doi: 10.1016/s1524-9042(02)54202-8. PMID 12836149
- [Background] Simavli S, Gumus I, Kaygusuz I, Yildirim M, Usluogullari B, Kafali H. Effect of music on labor pain relief, anxiety level and postpartum analgesic requirement: a randomized controlled clinical trial. Gynecol Obstet Invest. 2014;78(4):244-50. doi: 10.1159/000365085. Epub 2014 Sep 16. PMID 25227477
- [Background] Santivanez-Acosta R, Tapia-Lopez ELN, Santero M. Music Therapy in Pain and Anxiety Management during Labor: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2020 Oct 10;56(10):526. doi: 10.3390/medicina56100526. PMID 33050409
- [Background] Liu YH, Chang MY, Chen CH. Effects of music therapy on labour pain and anxiety in Taiwanese first-time mothers. J Clin Nurs. 2010 Apr;19(7-8):1065-72. doi: 10.1111/j.1365-2702.2009.03028.x. PMID 20492051
- [Background] Koch ME, Kain ZN, Ayoub C, Rosenbaum SH. The sedative and analgesic sparing effect of music. Anesthesiology. 1998 Aug;89(2):300-6. doi: 10.1097/00000542-199808000-00005. PMID 9710387
- [Background] Hosseini SE, Bagheri M, Honarparvaran N. Investigating the effect of music on labor pain and progress in the active stage of first labor. Eur Rev Med Pharmacol Sci. 2013 Jun;17(11):1479-87. PMID 23894767
- [Background] Fong TM, Drzymalski DM. The 95% Effective Duration of Music for Anxiolysis Before Elective Cesarean Delivery. A A Pract. 2025 Feb 28;19(3):e01931. doi: 10.1213/XAA.0000000000001931. eCollection 2025 Mar 1. PMID 40019185
- [Background] Drzymalski DM, Tsen LC, Palanisamy A, Zhou J, Huang CC, Kodali BS. A Randomized Controlled Trial of Music Use During Epidural Catheter Placement on Laboring Parturient Anxiety, Pain, and Satisfaction. Anesth Analg. 2017 Feb;124(2):542-547. doi: 10.1213/ANE.0000000000001656. PMID 27984250

DOCUMENTS (1):
  • Informed Consent Form (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT06969105/ICF_000.pdf